CLINICAL TRIAL: NCT05666310
Title: The Impact of Osteoporosis Medications on Muscle Health in Older Adults
Brief Title: Muscle Impact of Treating Osteoporosis
Acronym: MITO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nami Safai Haeri (Other)
Collaborators: The Claude D. Pepper Older Americans Independence Centers (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Nami Safai Haeri, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY22080139; P30AG024827 (NIH)
Record Dates: First submitted 2022-12-15; First posted 2022-12-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenia; Osteoporosis
MeSH Terms: conditions — Sarcopenia; Osteoporosis | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zoledronic Acid (Active Comparator)
  Interventions: Drug: Zoledronic Acid; Other: Denosumab Placebo
- Denosumab (Active Comparator)
  Interventions: Drug: Denosumab; Other: Zoledronic Acid Placebo

INTERVENTIONS:
Drug: Denosumab — Half of study participants will randomly receive denosumab 60 mg subcutaneous injection at month 0 and 6 with zoledronic acid placebo at month 0.
  Arms: Denosumab
Drug: Zoledronic Acid — Half of study participants will randomly receive zoledronic acid 5 mg intravenous infusion at month 0 with denosumab placebo at month 0 and 6. All forty participants will receive zoledronic acid 5 mg intravenous infusion at month 12.
  Arms: Zoledronic Acid
Other: Denosumab Placebo — Half of study participants who will randomly receive zoledronic acid 5 mg intravenous infusion at month 0 will also receive denosumab placebo at month 0 and 6.
  Arms: Zoledronic Acid
Other: Zoledronic Acid Placebo — Half of study participants who will randomly receive denosumab 60 mg subcutaneous injection at month 0 and 6 will also receive zoledronic acid placebo.
  Arms: Denosumab

SUMMARY:
Osteosarcopenia is a geriatric musculoskeletal syndrome characterized by co-existence of osteoporosis and sarcopenia (low skeletal muscle mass, strength, and/or functional capacity). There is strong evidence of overlap between the pathophysiology of osteoporosis and sarcopenia (muscle-bone crosstalk). This research plan will further explore the relationship between bone and muscle, and provide new information about effect of osteoporosis medications on muscle health in older adults who are under treatment for osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

Ambulatory adults age ≥65 years including those using assistive devices to maximize generalizability, if they have criteria for treating osteoporosis including:

1. Osteoporosis by axial bone density (spine, hip or forearm BMD T-score ≤-2.5 SD) or
2. A previous adult fragility fracture of the spine or hip or
3. Would be treated based on FRAX National Osteoporosis Foundation treatment thresholds of a 10-year risk of ≥ 20% for a major osteoporotic fracture or ≥ 3% for hip fracture using femoral neck BMD.

Exclusion Criteria:

1. Patients with a calculated creatinine clearance < 35 ml/min or
2. Who have a contraindication for bisphosphonates or denosumab or
3. Those who are scheduled for a tooth extraction to avoid jaw osteonecrosis or
4. Subjects with severe liver disease or
5. Those who have been on oral bisphosphonates for the past 1 year and intravenous bisphosphonates for the past 2 years prior to the study or
6. Men

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-14 (Actual); Primary Completion 2026-01-05 (Actual); Study Completion 2026-09-05 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in muscle mass (kg) measured by D3-Creatine | Baseline vs Month 12
  D3-Creatine dilution method is a novel method to measure muscle mass
Percentage change from baseline in appendicular lean mass (ALM/body mass index) | Baseline vs Month 12
  Appendicular lean mass is measured by whole body DXA scan and is an index of skeletal muscle mass
Percentage change from baseline in trabecular bone score (TBS) | Baseline vs Month 12
  TBS is measure of bone microarchitecture and is measured by a DXA system. A value of ≥ 1.35 indicates a normal architecture while TBS ≤ 1.20 indicates degraded microarchitecture
Percentage change from baseline in bone mineral density (BMD) (g/cm²) | Baseline vs Month 12
  BMD is measured by a DXA scan system and a higher BMD is correlated with lower fracture risk
Percentage change from baseline in grip strength (kgf) | Baseline vs Month 12
  Grip strength is measure of muscle strength and will be measured by a standard hand dynamometer
Percentage change from baseline in gait speed (m/s) | Baseline vs Month 12
  Gait speed is a measure of muscle function and will be measured by standard 4 meter gait speed test
Percentage change from baseline in rectus femoris muscle thickness (cm) | Baseline vs Month 12
  This variable will be measured by ultrasound
Percentage change from baseline in rectus femoris muscle cross-sectional surface area (cm²) | Baseline vs Month 12
  This variable will be measured by ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Nami Safai Haeri, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes

DOCUMENTS (1):
  • Informed Consent Form (2023-09-19): https://cdn.clinicaltrials.gov/large-docs/10/NCT05666310/ICF_000.pdf